CLINICAL TRIAL: NCT03519269
Title: Conventional vs. Robotic-Assisted Total Knee Arthroplasty: A Prospective, Randomized Trial of Clinical, Functional, and Radiographic Outcomes
Brief Title: Navio Robotic Versus Conventional Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Herbert John Cooper, MD, Assistant Professor of Orthopaedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR6537
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee replacement; robotic surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non robotics-assisted Surgical System (No Intervention): Conventional, non-robotics-assisted total knee surgical system
- Navio™ Robotics-assisted Surgical System (Experimental): Navio™ Robotics-assisted Surgical System
  Interventions: Device: Navio™ Robotics-assisted Surgical System

INTERVENTIONS:
Device: Navio™ Robotics-assisted Surgical System — Intervention will evaluate the utility of robotic-assistance in patients undergoing total knee arthroplasty
  Arms: Navio™ Robotics-assisted Surgical System

SUMMARY:
Total knee replacement surgery is a conventional approach to alleviating the pain and lack of function resulting from arthritis of the knee. While conventional knee replacement surgery is highly successful, incidences of improperly installed replacement parts are not uncommon. To improve outcomes, robotic-assisted total knee replacement surgery has recently become available, and has been shown to be extremely effective for partial knee replacement surgery. However, further research is needed to determine if this same technology can be equally effective for total knee replacement surgery. The present study will evaluate outcomes of robotic-assisted versus conventional total knee replacement surgery in patients between 40 and 85 years old with end stage arthritis of the knee. Other than surgical technique, patients will receive the same operative care and knee replacement implants. In addition to standard x-rays, subjects will be asked to complete several short-term clinical and functional tests and questionnaires to determine outcomes of their surgery.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) is a widespread orthopaedic procedure for restoring functionality and minimizing pain due to end stage osteoarthritis. Conventional TKA, well-accepted as the standard of care, is performed with manual instrumentation guided by intramedullary or extramedullary alignment rods, as well as rotational guides that are not patient-specific. Despite continued improvement in manual instrumentation, postoperative malalignment is still reported in a significant number of patients when these manual instruments are used. Robotic-assisted TKA was developed specifically to improve surgical accuracy, and has been shown to significantly improve accuracy of alignment and joint-line restoration. However, these improvements came at the cost of higher complication rates and were not shown to translate into meaningful clinical outcomes with these first-generation systems. Newer-generation robotic technology offers several advantages over earlier versions including the potential to dynamically assess soft tissues over a range of motion and the ability to use haptic control in bone preparation. Modern robotic-assisted knee surgery has also demonstrated superior outcomes over conventional instrumentation in unicompartmental knee arthroplasty (UKA). This newer-generation of robotic technology, which has quickly become the standard-of-care for many knee surgeons who perform UKA, has recently been approved by the United States Food and Drug Administration (FDA) for use in TKA. Prior to consideration of widespread adoption of this newer technology in patients undergoing TKA, well-designed clinical trials are necessary to study its efficacy in this population. The proposed study evaluates the efficacy of robotic-assistance in patients between 40 and 85 years old with end-stage knee osteoarthritis or degenerative joint disease undergoing TKA. It is designed as a prospective, randomized trial where patients are blinded to their treatment arm. Patients will be randomized to conventional vs. robotically-assisted techniques in the operating room and, other than the surgical technique, will receive the same perioperative care and identical implants. The investigators aim to measure utility of robotic-assisted TKA through a range of early and short-term clinical, functional, and radiographic outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 85
* body mass index (BMI) less than 40.0 kg/m^2
* end-stage knee osteoarthritis (Kellgren and Lawrence grade 4)
* failure of a minimum 12 weeks of nonoperative management
* English fluency

Exclusion Criteria:

* history of inflammatory arthropathy in the same knee
* history of prior open knee surgery in the same knee
* history of prior osteotomy or periarticular fracture
* deformity > 15 degrees from a neutral mechanical axis
* gross ligamentous incompetence of the medial or lateral collateral ligaments
* musculoskeletal involvement beyond unilateral knee osteoarthritis significantly limiting their function
* unwillingness or inability to participate in the proposed study protocol and follow-up

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Score on Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Up to 2 years
  The WOMAC is a 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function. Scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Score on the Timed Up and Go Test (TUG) | Up to 2 years
  The TUG measures the time (in seconds) it takes a patient to rise from an armed chair, walk 3 meters, turn, and return to sitting in the same chair. The time taken to complete the task is strongly correlated to level of functional mobility, (i.e., the more time taken, the more dependent in activities of daily living). Risk for Falls: high risk (>13.5 seconds), none/low/moderate (<13.5 seconds).

SECONDARY OUTCOMES:
Score on Short-Form 12 Health Questionnaire (SF-12) | Up to 2 years
  The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. Questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Score on New Knee Society Scores (2011 KSS) | Up to 2 years
  The 2011 KSS is a physician- and patient-derived scoring system that has been validated and demonstrated to be a responsive method for assessing objective and subjective outcomes after TKA. This scale comprises four separate subscales: (a) objective knee score (seven items: 100 points); (b) patient satisfaction score (five items: 40 points); (c) patient expectations score (three items: 15 points); and (d) functional activity score (19 items: 100 points). Score 80-100: Excellent; Score 70-79: Good; Score 60-69: Fair; Score below 60: Poor
Score on Global Rating Score of Knee Function (GRS) | Up to 2 years
  Participants will be asked to rate their perception of knee functional ability on a scale of 0 to 100%. A score of 0 represents a complete disability and a score of 100 represents a level of knee function prior to the patient having any symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert John Cooper, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No